CLINICAL TRIAL: NCT06044922
Title: Heart Rate Variability in Early Prediction of a Noxic Brain Injury After Cardiac Arrest
Acronym: HEAVENwARd
Status: Recruiting | Type: Observational
Sponsor: CMC Ambroise Paré (Other)
Responsible Party: Sponsor
Other Study IDs: 2022/01
Record Dates: First submitted 2023-09-13; First posted 2023-09-21 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Cardiac Arrest
Keywords: Heart rate variability; Neurologic prognosis
MeSH Terms: conditions — Heart Arrest | interventions — Electrocardiography, Ambulatory

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Post-cardiac arrest patients
  Interventions: Device: 24-hour Holter monitoring

INTERVENTIONS:
Device: 24-hour Holter monitoring — Holter monitor is fitted within 2h of ICU admission to acquire a 24-hour electrocardiogram recording

SUMMARY:
Despite advances in post-resuscitation care of patients with cardiac arrest (CA), the majority of survivors who are treated after restoration of spontaneous circulation (ROSC) will have sequelae of hypoxic-ischemic brain injury ranging from mild cognitive impairment to a vegetative state.

Early prognostication in comatose patients after ROSC remains challenging. Recent recommendations suggest carrying out clinical and paraclinical tests during the first 72 h after ROSC, to predict a poor neurological outcome with a specificity greater than 95% (no pupillary and corneal reflexes, bilaterally absent N20 somatosensory evoked potential wave, status myoclonus, highly malignant electroencephalography including suppressed background ± periodic discharges or burst-suppression, neuron-specific enolase (NSE) > 60 µg/L, a diffuse and extensive anoxic injury on brain CT/MRI), but with a low sensitivity due to frequent confounding factors.

The heart rate variability (HRV) is a simple and non-invasive technique for assessing the autonomic nervous system function. In patients with a recent myocardial infarction, reduced HRV is associated with an increased risk for malignant arrhythmias or death. In neurology, reduced HRV is associated with a poor outcome in severe brain injury patients and allows to predict early neurological deterioration and recurrent ischemic stroke after acute ischemic stroke.

A reduced HRV could be a sensitive, specific and early indicator of diffuse anoxic brain injury after CA.

This multicenter prospective cohort study assesses the added value of early HRV (within 24h of ICU admission) for neuroprognostication after cardiac arrest.

ELIGIBILITY:
Inclusion Criteria:

* Admitted in intensive care unit (ICU) after resuscitation from cardiac arrest (in-hospital or out-of-hospital)
* Coma (Glasgow score < 8) after ROSC, requiring sedation and targeted temperature management for at least 24h

Exclusion Criteria:

* Dying patient (Limitation of life support techniques at admission to the ICU)
* Non-Sinus Rhythm
* Pregnant or breastfeeding women
* Patient under protection of the adults (guardianship, curators or safeguard of justice)
* Opposition by the trusted person or by the patient once he/she wakes up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Comatose patients admitted in ICU after resuscitation from cardiac arrest
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-10-23 (Actual); Primary Completion 2027-12-15 (Estimated); Study Completion 2027-12-15 (Estimated)

PRIMARY OUTCOMES:
Poor neurological outcome evaluated using the CPC score | At day-28
  The CPC (Cerebral Performance Category) score assesses neurological status after cardiac arrest on a scale of 1 to 5 (1 = conscious and normal; 2 = conscious with moderate disability; 3 = conscious with severe disability; 4 = coma or vegetative state; 5 = death).
  The CPC score will be dichotomized as follow: good neurological outcome for categories 1 and 2 and poor neurological outcome or death for categories 3, 4 and 5.
  The CPC score will be obtained at day-28 from an in-hospital visit if the patient is still hospitalized or by phone call if patient returned home.

SECONDARY OUTCOMES:
Net reclassification index | At day-28
Brain death | At day-28
Days without limitation of life sustaining treatment | At day-28

CONTACTS AND LOCATIONS:
Locations (5):
- France (5):
  - Brest University Hospital, Brest, Brittany Region
  - Nantes University Hospital, Nantes, Pays de la Loire Region
  - Marseille University Hospital, Marseille, Provence-Alpes-Côte d'Azur Region
  - Ambroise Paré - Hartmann Private Hospital Group, Neuilly-sur-Seine, Île-de-France Region
  - Cochin Hospital, Paris, Île-de-France Region

IPD SHARING:
Plan to Share IPD: No